CLINICAL TRIAL: NCT04280263
Title: A Prospective Double Blinded Randomized Placebo Controlled Study of the Efficacy of Caffeine as an Analgesic Adjuvant for Acute Perioperative Pain Management Following Total Joint Arthroplasty
Brief Title: Caffeine Study for Pain Control Following Total Joint Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020 DP
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffiene (Active Comparator): This group will receive 150mg caffeine tablets to be taken twice per day
  Interventions: Drug: Caffeine
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Caffeine — caffeine tables containing 150mg caffeine will be provided to patients with instructions to take twice per day
  Arms: Caffiene
Drug: Placebo oral tablet — oral placebo tablets matching the caffeine tablets and will be provided to patients with instructions to take twice per day
  Arms: placebo

SUMMARY:
A prospective, double blinded, single center, randomized controlled study to evaluate the efficacy of caffeine in combination with acetyl salicylic acid (ASA) in the management of postoperative pain in patients undergoing total joint arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patient is older than 18 years old at the time of the surgery.
* Patient is treated by Rothman Orthopaedics institute and is scheduled for the surgical procedure at AtlantiCare Regional Medical Center.
* Patient is undergoing total hip or total knee arthroplasty.
* Patient has the diagnosis of Osteoarthritis of the hip or the knee, or other noninflammatory disease that results in joint damage to the hip or the knee.

Exclusion Criteria:

* Patient has known history of opioid addiction and/or has taken opioids preoperatively.
* Patient has history of cardiac diseases that might be aggravated by the use of caffeine, as diagnosed by a cardiologist or demonstrated by an abnormal EKG.
* Patient has a known allergy to aspirin or caffeine.
* Patient has history of chronic pain that required the intervention of a pain management doctor.
* Patient has an active infection at the time of surgery (systemic or localized) or history of chronic infections that affected the lower extremities.
* Patient has history of cancer that would affect patient reported outcomes including pain.
* Patient has history of neuropathic pain or nerve degenerative disease.
* Patients undergoing revision surgery would be excluded.
* Patients who require alternate DTV prophylaxis other than ASA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
post-operative pain | 2 weeks post-operative
  pain will be recorded via Visual Analog Scale (VAS). The scale ranges from zero to 100 with zero being no pain and 100 being worst pain imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedics at Egg Harbor Township, Egg Harbor, New Jersey, United States